CLINICAL TRIAL: NCT00159146
Title: A Short Term Double Blind Randomised Trial of Pindolol Augmentation in Venlafaxine Treated Patients With Major Depression
Brief Title: Trial of Pindolol Augmentation in Venlafaxine Treated Patients With Major Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of participants fulfilling inclusion criteria
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Tvergaards Foundation (Unknown)
Responsible Party: Klaus Martiny, Psychiatric Research Unit, Hillerod Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: version 5
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Major Depression
Keywords: Major Depression; Pindolol; Venlafaxine; Augmentation; Major depression (DSM-IVR)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Pindolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Venlafaxine and pindolol
  Interventions: Drug: Pindolol and venlafaxin
- B (Placebo Comparator): Venlafaxin and placebo
  Interventions: Drug: Pindolol and venlafaxin

INTERVENTIONS:
Drug: Pindolol and venlafaxin — pindolol 20 mg and venlafaxin 150 mg

SUMMARY:
This study investigates the hypothesis that pindolol can accelerate the response to antidepressants in patients with major depression treated with venlafaxine.

DETAILED DESCRIPTION:
Antidepressant therapy has a delayed onset of action of 4-6 weeks. Pindolol has in some studies shown an accelerating effect. In this study we investigate the effect of 20 mg of pindolol retarded formulation in combination with Venlafaxine compared to placebo Pindolol and Venlafaxine for a duration of 19 days.

Effect is measured by the Hamilton Depression rating Scale and the Preskorn Scale (self-rating).

ELIGIBILITY:
Inclusion Criteria:

* Major depression

Exclusion Criteria:

* Allergy towards pindolol, venlafaxine or other tablet constituents
* Liver or kidney impairment
* Diabetics
* Age below 18 years
* Severe cardiac disease
* Asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale scores | 1 week

SECONDARY OUTCOMES:
Preskorn scores | one day

CONTACTS AND LOCATIONS:
Overall Officials: Per Bech, Professor, Study Chair — Psychiatric Research Unit, Hillerod Hospital
Locations (1):
- Psychiatric Research Unit, Hillerod Hospital, Hillerød, Denmark

REFERENCES:
- [Derived] Martiny K, Lunde M, Bech P, Plenge P. A short-term double-blind randomized controlled pilot trial with active or placebo pindolol in patients treated with venlafaxine for major depression. Nord J Psychiatry. 2012 Jun;66(3):147-54. doi: 10.3109/08039488.2012.674553. Epub 2012 Mar 29. PMID 22458638